CLINICAL TRIAL: NCT04444830
Title: Can Intranasal Ketorolac Tromethamine Prescribed Postoperatively After Major Female Pelvic Reconstructive Surgery Reduce Consumption of Prescribed Narcotics?
Brief Title: Sprix for Postoperative Pain Control Following Gynecologic Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study never opened to enrollment. Study never IRB approved.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Sean Francis, MD, Chairperson & Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.1351
Record Dates: First submitted 2020-06-07; First posted 2020-06-24 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain Control; Narcotic Use; Pelvic Organ Prolapse; Urinary Incontinence , Stress; Surgery
Keywords: Minimally Invasive Gynecologic Surgery; Female Pelvic Reconstructive Surgery; Post Operative Pain Control; Narcotic Reduction; Opioid Reduction; Pelvic Organ Prolapse; Stress Urinary Incontinence
MeSH Terms: conditions — Pelvic Organ Prolapse; Urinary Incontinence, Stress | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: This is a multi-center, non-blinded, randomized control trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard (No Intervention): To compare the total amount of opioid consumption, as measured by morphine mEq, consumed in patients immediately postoperative from minimally invasive female pelvic reconstructive surgery - they will be prescribed a "standard" postoperative regimen of Acetaminophen 650 mg PO q 6-8 hours + Ibuprofen 600 mg PO q 6-8 hours + rescue narcotics (Oxycodone 5-10 mg PO q 4-6 hours or if allergic to Oxycodone, Norco 5-10mg/325mg PO q 4-6 hours) for breakthrough pain
- Sprix (Experimental): To compare the total amount of opioid consumption, as measured by morphine mEq, consumed in patients immediately postoperative from minimally invasive female pelvic reconstructive surgery - they will be prescribed regimen of Sprix 30.5mg Intranasal q 6-8 hour up to 4 times daily + Acetaminophen 650 mg PO q 6- 8 hours + rescue narcotics (as above) for breakthrough pain during the day of surgery and the following 4 postoperative days.
  Interventions: Drug: Sprix

INTERVENTIONS:
Drug: Sprix — Intranasal Ketorolac - used as directed for an appropriate, previously established indication
  Other Names: Intranasal Ketorolac
  Arms: Sprix

SUMMARY:
The ongoing opioid epidemic has altered both how physicians prescribe narcotics and patients' perceptions of those prescriptions. Along with increased scrutiny regarding the quantity of opioids that be may prescribed after acute injury, for chronic conditions and following surgery the healthcare industry as a whole continues to search for alternative medications that provide adequate pain relief and have a reduced tendency for abuse/dependence/addition. To that end this study has the following aims:

1. To evaluate the amount of opioids consumed following minimally invasive, female pelvic surgery when patients' postoperative pain is managed via:

   1. Acetaminophen plus Ibuprofen plus breakthrough pain opioids (Standard protocol)
   2. Acetaminophen plus Intranasal Ketorolac Tromethamine plus opioids for breakthrough pain (Sprix protocol)
2. Patient satisfaction with the aforementioned methods
3. Evaluate and compare pain scores via validated questionnaire

Hypothesis:

Primary:

1. Patients prescribed intranasal Ketorolac (Sprix protocol) will consume significantly less Morphine Milliequivalents (mEqs) of narcotics compared to the standard protocol following minimally invasive female pelvic surgery.

Secondary:

1. Patients in the Sprix protocol will have lower Visual Analog Scale (VAS) measures of pain which will be measured on a 0-10 scale where 0 denotes no pain and 10 denotes maximum experience of pain
2. Patients in the Sprix protocol will have lower numeric pain score and on POD#4
3. Patients in the Sprix protocol will have higher Quality of Recovery 40 (QoR-40 )scores on POD#1
4. Patients in the Sprix protocol will have higher QoR-40 scores on POD#4
5. Patients will not have any significant difference in overall surgical satisfaction on POD#1 and POD#4 using a numerical satisfaction score
6. Patients in the Sprix protocol will be more likely to consume no narcotics at all once discharged to home

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age
2. Weight ≥ 110lbs
3. English Speaking and Reading
4. All consecutive, consenting female patients undergoing Pelvic Organ Prolapse (POP) surgery - vaginal prolapse surgery, laparoscopic vaginal prolapse surgery or robotic assisted vaginal prolapse surgery - with or without Bilateral or Unilateral Salpingoopherectomy, with or without concomitant hysterectomy, with or without urinary anti-incontinence surgery

Exclusion Criteria:

1. Patients taking opioids chronically at the time of surgery
2. History of Coronary Artery Bypass Graft (CABG)
3. History of peptic ulcer disease or bleeding in the stomach or intestines
4. History of asthma attack, hives, or other allergic reaction with aspirin or any other Non-Steroidal Anti-inflammatory Drug (NSAID)
5. Uncontrolled hypertension at the time of consent and/or surgery
6. History of renal impairment as defined by blood creatinine of 1.1 or greater at any time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients - all patients in the study are those that will undergo/have undergone female pelvic surgery (Urogynecology)
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Morphine mEqs | As measured from the day of surgery to 4 days post operative
  The amount of narcotics consumed postoperatively as measure by Morphine milliequivalents

SECONDARY OUTCOMES:
Patient Satisfaction | Day of surgery to 4 days postoperative
  Evaluate patient satisfaction using the validated QoR 40 (Quality of Recovery) Scale - wherein a minimum score of 40 indicates that a patient perceives there recovery to be very poor and a maximum score of 200 indicates that the patient perceives that the quality of their recovery is excellent
Patient's perception of current pain | Day of surgery to 4 days postoperatively
  The patient's pain will be subjectively scaled on a 0 (indicating no pain) to 10 (indicating maximum/severe pain) scale. The patient will be asked to scale their pain preoperatively, on postoperative day #1 and on Postoperative day #4

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singla N, Singla S, Minkowitz HS, Moodie J, Brown C. Intranasal ketorolac for acute postoperative pain. Curr Med Res Opin. 2010 Aug;26(8):1915-23. doi: 10.1185/03007995.2010.495564. PMID 20557145
- [Background] Pergolizzi JV Jr, Taylor R Jr, Raffa RB. Intranasal ketorolac as part of a multimodal approach to postoperative pain. Pain Pract. 2015 Apr;15(4):378-88. doi: 10.1111/papr.12239. Epub 2014 Aug 28. PMID 25169467
- [Background] Pollack CV Jr, Diercks DB, Thomas SH, Shapiro NI, Fanikos J, Mace SE, Rafique Z, Todd KH. Patient-reported Outcomes from A National, Prospective, Observational Study of Emergency Department Acute Pain Management With an Intranasal Nonsteroidal Anti-inflammatory Drug, Opioids, or Both. Acad Emerg Med. 2016 Mar;23(3):331-41. doi: 10.1111/acem.12902. PMID 26782787
- [Background] Moodie JE, Brown CR, Bisley EJ, Weber HU, Bynum L. The safety and analgesic efficacy of intranasal ketorolac in patients with postoperative pain. Anesth Analg. 2008 Dec;107(6):2025-31. doi: 10.1213/ane.0b013e318188b736. PMID 19020154